CLINICAL TRIAL: NCT01542073
Title: 68Ga-BNOTA-PRGD2 PET/CT in Evaluation of Angiogenesis of Myocardial Infarction and the Comparison With Cardiac Perfusion and Metabolism
Brief Title: 68Ga-BNOTA-PRGD2 PET/CT in Evaluation of Myocardial Infarction
Acronym: GRGDMI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM003
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
Keywords: myocardial infarction; angiogenesis; integrin receptor imaging; 68Ga-BNOTA-PRGD2
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — 68gallium-BNOTA-PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BNOTA-PRGD2 cardiac PET/CT scanning (Experimental): We will perform 68Ga-BNOTA-PRGD2 cardiac PET/CT scanning on myocardial infarction patients to determine its value.
  Interventions: Drug: 68Ga-BNOTA-PRGD2

INTERVENTIONS:
Drug: 68Ga-BNOTA-PRGD2 — Intravenous injection of one dosage of 111 MBq 68Ga-BNOTA-PRGD2. Tracer doses of 68Ga-BNOTA-PRGD2 will be used to image angiogenesis of myocardial infarction area by positron emission tomography / computed tomography (PET/CT)
  Other Names: 68Ga-p-SCN-Bn-NOTA-PEG3-RGD2

SUMMARY:
This is an open-label PET/CT (positron emission tomography/computed tomography) study to investigate the diagnostic performance of 68Ga-BNOTA-PRGD2 in evaluation of myocardial infarction. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into myocardial infarction patients. Visual and semiquantitative method will be used to assess the 68Ga-BNOTA-PRGD2 PET/CT cardiac images and compared to the 99mTc-MIBI SPECT myocardial perfusion images and the 18F-FDG metabolism images.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of integrin receptor family and expressed preferentially on regenerative vascular endothelial cells and some tumor cells, but not or very low expressed on the quiescent vessel cells and other normal cells. The αvβ3 integrin is a key mediator of angiogenesis and thus may be an important diagnostic and therapeutic target associated with myocardial repair processes after ischaemic injury.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 expression via positron emission tomography (PET) or single photon emission computed tomography (SPECT). Among all the RGD radiotracers studied in Myocardial Infarction (MI), 18F-Galacto-RGD and 99mTc-RGD has been investigated clinically in acute MI patients, showing focal tracer retention localized in the infarcted area. Recently, series of RGD dimeric peptides with PEG linkers have been developed. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence. As a representative, 68Ga-BNOTA-PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in both animal and human studies to date.

For the further interests in clinical translation of 68Ga-BNOTA-PRGD2, a open-label PET/CT study was designed to investigate the diagnostic performance of 68Ga-BNOTA-PRGD2 in myocardial infarction patients. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 ( ≤ 40 µg BNOTA-PRGD2) will be intravenously injected into the myocardial infarction patients. Visual and semiquantitative method will be used to assess the PET/CT images. 99mTc-MIBI myocardial perfusion SPECT images and 18F-FDG metabolism images will be used for co-registrated comparison.

ELIGIBILITY:
Inclusion Criteria:

Myocardial infarction patients:

* Males and females
* ≥30 years old
* Patients had myocardial infarction diagnosis (fulfilling two or three symptoms: clinical history of ischaemic type chest pain lasting for more than 20 minutes, changes in serial ECG tracings, rise and fall of serum cardiac biomarkers such as creatine kinase-MB fraction and troponin)

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Have other kinds of heart diseases
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment (Standardized Uptake Values = SUVs) of myocardial infarction region and normal left ventricular wall | 1 year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician and will compare to 99mTc-MIBI myocardial perfusion imaging and 18F-FDG myocardial metabolism imaging obtained within a week. The semiquantitative analysis will be performed by the same person for all the cases, and the MI region standardized uptake values (SUVs), the SUV ratios (SUV of MI/SUV normal LV), and other organs' SUVs will be measured.

SECONDARY OUTCOMES:
Number of participants with adverse events | 1 year
  Adverse events within 5 days after 68Ga-BNOTA-PRGD2 injection and PET/CT scanning of the patients will be collected and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Department of Nuclear Medicine, Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No